CLINICAL TRIAL: NCT02347527
Title: Neuronal and Behavioral Effects of Implicit Priming in Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-1786; R21DK102052 (NIH); P30DK048520 (NIH)
Record Dates: First submitted 2015-01-16; First posted 2015-01-27 (Estimated); Results first posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Feeding Behavior; Obesity; Overweight
MeSH Terms: conditions — Feeding Behavior; Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: The "MRI sample" and "Behavioral-only sample" involve separate participants who complete the same intervention (assigned to either active or control groups), but the "MRI sample" also completed MRI outcomes and a food intake outcome that the "Behavioral-only sample" did not.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active Implicit Priming (MRI sample) (Experimental): Participants will complete active implicit priming, in which food images are implicitly primed (i.e., below conscious awareness) with images of positive or negative affect. In addition to measures of food image ratings, this group completed a visual food cues scan during fMRI to assess change in neuronal response to food cues. They also completed a measure of food intake post-intervention.
  Interventions: Behavioral: Active Implicit Priming
- Control Implicit Priming (MRI sample) (Placebo Comparator): Participants will complete a control implicit priming intervention, which matches the active intervention, but with neutral stimuli as primes. In addition to measures of food image ratings, this group completed a visual food cues scan during fMRI to assess change in neuronal response to food cues. They also completed a measure of food intake post-intervention.
  Interventions: Behavioral: Control Implicit Priming
- Active Implicit Priming (Behavioral-only sample) (Experimental): Participants will complete active implicit priming, in which food images are implicitly primed (i.e., below conscious awareness) with images of positive or negative affect.
  Interventions: Behavioral: Active Implicit Priming
- Control Implicit Priming (Behavioral-only sample) (Placebo Comparator): Participants will complete a control implicit priming intervention, which matches the active intervention, but with neutral stimuli as primes.
  Interventions: Behavioral: Control Implicit Priming

INTERVENTIONS:
Behavioral: Active Implicit Priming — A 10-minute implicit priming intervention, associating food images with images of positive or negative valence.
  Arms: Active Implicit Priming (Behavioral-only sample); Active Implicit Priming (MRI sample)
Behavioral: Control Implicit Priming — A 10-minute implicit priming intervention, associating food images with images of neutral valence.
  Arms: Control Implicit Priming (Behavioral-only sample); Control Implicit Priming (MRI sample)

SUMMARY:
The overall goals of this project are to determine the impact of an implicit priming intervention, designed to alter food perceptions, on both brain responses to food and on food intake behaviors in overweight/obese individuals. The investigators hypothesized that this bottom-up sensory-level conditioning approach would effectively result in reduced preference for high-calorie foods.

DETAILED DESCRIPTION:
One factor that may contribute to susceptibility to obesity is a high responsivity to high-calorie foods in terms of cognitive factors such as emotional associations, reward value or reinforcing properties of food. Many of these processes involve learned associations thought to develop via classical conditioning through repeated pairings with external stimuli, which can influence food preferences and intake. As such, improving our understanding of the neuronal mechanisms underlying these processes and attempting to modify them may be a useful strategy to promote weight loss and maintenance. Therefore, the proposed study aims to investigate the effects of altering food perception on neuronal responses and food intake behaviors by using implicit priming, in which positively or negatively valenced images are presented immediately prior to food images, but are not consciously perceived.

The project goals are to determine the impact of the implicit priming intervention on both brain responses to food cues and on food intake behaviors in overweight/obese individuals. Food image ratings were assessed before and after either (a) an active implicit priming intervention or (b) a control intervention. One group of participants (n = 47; "MRI sample") completed the intervention during an fMRI scan and completed a visual food cues task both before and after the intervention (during fMRI), to assess intervention-related change in neuronal responses to food cues. In this group, food intake measures were also taken following fMRI. In a separate group of participants (n = 45; "Behavioral-only sample"), the primary outcome measure was the change in food image ratings from pre- to post-intervention; fMRI and measures of food intake were not assessed in this group.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese adults
* Healthy weight adults

Exclusion Criteria:

* Vegetarian, vegan, or having other wide-ranging food restrictions
* Currently dieting
* MRI exclusion criteria, if in MRI sample (e.g., claustrophobia, metal in the body)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason R Tregellas, PhD, Principal Investigator — University of Colorado, Denver; Kristina T Legget, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Legget KT, Cornier MA, Erpelding C, Lawful BP, Bear JJ, Kronberg E, Tregellas JR. An implicit priming intervention alters brain and behavioral responses to high-calorie foods: a randomized controlled study. Am J Clin Nutr. 2022 Apr 1;115(4):1194-1204. doi: 10.1093/ajcn/nqac009. PMID 35030242
- [Derived] Legget KT, Cornier MA, Rojas DC, Lawful B, Tregellas JR. Harnessing the power of disgust: a randomized trial to reduce high-calorie food appeal through implicit priming. Am J Clin Nutr. 2015 Aug;102(2):249-55. doi: 10.3945/ajcn.115.106955. Epub 2015 Jun 24. PMID 26109580

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the "Behavioral-Only" sample, participants were recruited via flyer advertisement in Aurora, CO, between May 2013 and March 2014. For the "MRI" sample, participants were recruited via email and flyer advertisement in Aurora, CO, between May 2015 and August 2019.
Pre-assignment Details: 47 participants were in the "MRI sample" and 45 were in the "Behavioral-only sample," for a total of 92 unique study participants.
Groups:
- Active Implicit Priming (MRI Sample): Participants completed active implicit priming, in which food images were implicitly primed (i.e., below conscious awareness) with images of positive or negative affect. This group completed the priming intervention during fMRI scanning.
  Active Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of positive or negative valence.
- Control Implicit Priming (MRI Sample): Participants completed a control implicit priming intervention, which matched the active intervention, but with neutral stimuli as primes. This group completed the priming intervention during fMRI scanning.
  Control Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of neutral valence.
- Active Implicit Priming (Behavioral-only Sample); Control Implicit Priming (Behavioral-only Sample): Participants completed active implicit priming, in which food images were implicitly primed (i.e., below conscious awareness) with images of positive or negative affect.
  Active Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of positive or negative valence.
Period: Overall Study
Arm/Group | Active Implicit Priming (MRI Sample) | Control Implicit Priming (MRI Sample) | Active Implicit Priming (Behavioral-only Sample) | Control Implicit Priming (Behavioral-only Sample)
Started | 25 | 22 | 23 | 22
Completed Intervention | 24 | 21 | 23 | 22
Included in Analyses | 22 | 19 | 22 | 20
Completed | 22 | 19 | 22 | 20
Not Completed | 3 | 3 | 1 | 2
Not completed — MRI not completed due to technical difficulties | 1 | 0 | 0 | 0
Not completed — MRI stopped due to participant anxiety | 0 | 1 | 0 | 0
Not completed — Excluded from analyses due to excess movement during MRI scan | 1 | 1 | 0 | 0
Not completed — Excluded from analyses due to technical difficulties during the study visit | 1 | 0 | 1 | 2
Not completed — Excluded from analyses due to non-compliance with study procedures | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Implicit Priming (MRI Sample): Participants completed active implicit priming, in which food images were implicitly primed (i.e., below conscious awareness) with images of positive or negative affect. This group completed the intervention during fMRI scan.
  Active Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of positive or negative valence.
- Control Implicit Priming (MRI Sample): Participants completed a control implicit priming intervention, which matched the active intervention, but with neutral stimuli as primes. This group completed the intervention during fMRI scan.
  Control Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of neutral valence.
- Control Implicit Priming (Behavioral-only Sample): Participants completed a control implicit priming intervention, which matched the active intervention, but with neutral stimuli as primes.
  Control Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of neutral valence.
- Total: Total of all reporting groups
Arm/Group | Active Implicit Priming (MRI Sample) | Control Implicit Priming (MRI Sample) | Active Implicit Priming (Behavioral-only Sample) | Control Implicit Priming (Behavioral-only Sample) | Total
Number analyzed (Participants) | 22 | 19 | 22 | 20 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (14.4) | 37.3 (13.6) | 30.7 (6.0) | 35.1 (11.88) | 36.15 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 14 | 12 | 54
  Male | 4 | 9 | 8 | 8 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 3 | 4 | 13
  Not Hispanic or Latino | 9 | 8 | 19 | 16 | 52
  Unknown or Not Reported | 8 | 10 | 0 | 0 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 2 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 1 | 3
  White | 16 | 13 | 17 | 14 | 60
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 3 | 4 | 14
Region of Enrollment [Number; unit: participants]
  United States | 22 | 19 | 22 | 20 | 41
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.8 (5.5) | 28.8 (3.0) | 22.5 (3.0) | 24.2 (4.4) | 29.8 (4.6)
Baseline food image ratings [Mean (Standard Deviation); unit: units on a scale] — Baseline ratings of high-calorie food cues on "desire to eat" (scale of 0-100, with higher numbers indicating higher desire to eat). Population: Due to technical difficulties, food cue ratings were not collected for 5 participants in the MRI sample groups (sample size for this measure for the MRI sample groups: active, n = 19; control n = 17).
  units on a scale
    number analyzed (Participants) | 19 | 17 | 22 | 20 | 78
    (all) | 62.2 (16.0) | 52.5 (14.3) | 54.8 (13.1) | 50.2 (22.5) | 55.1 (14.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Food Image Ratings
Description: Food image ratings (high-calorie foods) change from baseline, measured within 10 minutes post-intervention. Food images are rated on "desire to eat" by visual analogue scale (0-100; higher scores mean greater desire to eat). Negative values indicate reduced scores post-intervention compared to baseline, with greater numbers indicating greater reduction.
Time Frame: Baseline to within 10 minutes post-intervention
Measure: Mean (Standard Error); unit: Score change from baseline
Groups:
- Active Implicit Priming (MRI Sample): Participants completed active implicit priming, in which food images were implicitly primed (i.e., below conscious awareness) with images of positive or negative affect. This group completed the intervention during an fMRI scan.
  Active Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of positive or negative valence.
- Control Implicit Priming (MRI Sample): Participants completed a control implicit priming intervention, which matched the active intervention, but with neutral stimuli as primes.This group completed the intervention during an fMRI scan.
  Control Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of neutral valence.
Arm/Group | Active Implicit Priming (MRI Sample) | Control Implicit Priming (MRI Sample) | Active Implicit Priming (Behavioral-only Sample) | Control Implicit Priming (Behavioral-only Sample)
Number analyzed (Participants) | 19 | 17 | 22 | 20
Score change from baseline | -5.1 (2.5) | -.3 (2.2) | -6.8 (1.3) | -2.7 (1.4)
Statistical Analysis 1: Comparison: Active Implicit Priming (MRI Sample) vs Control Implicit Priming (MRI Sample); Test type: Superiority; p = 0.038, ANOVA
Statistical Analysis 2: Comparison: Active Implicit Priming (Behavioral-only Sample) vs Control Implicit Priming (Behavioral-only Sample); Test type: Superiority; p = 0.036, ANOVA

2. Primary Outcome: Neuronal Response to Food Cues
Description: Neuronal response while viewing visual food cues will be measured using functional magnetic resonance imaging (fMRI). Primary outcome was insula response change from baseline, as measured within 20 minutes after the intervention. A bilateral region of interest (ROI) for the insula was defined anatomically, with mean difference from baseline to post-intervention (% BOLD signal change) calculated across all voxels for that ROI. A positive number indicates a reduced response (with higher numbers indicating greater change) and a negative number indicates an increased response.
Time Frame: Baseline to post-intervention
Measure: Mean (Standard Deviation); unit: % BOLD signal change from baseline
Groups:
- Active Implicit Priming: Participants completed active implicit priming, in which food images were implicitly primed (i.e., below conscious awareness) with images of positive or negative affect.
  Active Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of positive or negative valence.
- Control Implicit Priming: Participants completed a control implicit priming intervention, which matched the active intervention, but with neutral stimuli as primes.
  Control Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of neutral valence.
Arm/Group | Active Implicit Priming | Control Implicit Priming
Number analyzed (Participants) | 21 | 19
% BOLD signal change from baseline | 0.21 (0.45) | -0.07 (.34)
Statistical Analysis 1: Comparison: Active Implicit Priming vs Control Implicit Priming; Test type: Superiority; p = 0.010, t-test, 2 sided

3. Secondary Outcome: Food Intake
Description: Food intake during ad-lib lunch (kcals)
Time Frame: 1 hour post-intervention
Measure: Mean (Standard Deviation); unit: kcals
Arm/Group | Active Implicit Priming | Control Implicit Priming
Number analyzed (Participants) | 19 | 17
kcals | 959.03 (343.53) | 860.38 (361.99)
Statistical Analysis 1: Comparison: Active Implicit Priming; Relationship between change in high-calorie food ratings and subsequent food intake (kcals); Test type: Other; p = 0.040, Pearson's correlation
Statistical Analysis 2: Comparison: Control Implicit Priming; Relationship between change in high-calorie food ratings and subsequent food intake (kcals); Test type: Other; p = 0.92, Pearson's correlation

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the one-day study day period.
Description: Occurrence of adverse events was assessed on an ongoing, case-by-case basis.
Groups:
- Active Implicit Priming (MRI Sample): Participants completed active implicit priming, in which food images were implicitly primed (i.e., below conscious awareness) with images of positive or negative affect. Participants in this group completed the intervention during an fMRI scan.
  Active Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of positive or negative valence.
- Control Implicit Priming (MRI Sample): Participants completed a control implicit priming intervention, which matched the active intervention, but with neutral stimuli as primes. Participants in this group completed the intervention during an fMRI scan.
  Control Implicit Priming: A 10-minute implicit priming intervention, associating food images with images of neutral valence.
Arm/Group | Active Implicit Priming (MRI Sample) | Control Implicit Priming (MRI Sample) | Active Implicit Priming (Behavioral-only Sample) | Control Implicit Priming (Behavioral-only Sample)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/19 | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/19 | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT02347527/Prot_SAP_000.pdf